CLINICAL TRIAL: NCT04067063
Title: Massive Mental Health Screening Using Smartphone in Milpa Alta Community, Mexico.
Brief Title: Population Screening Using Smartphone in Milpa Alta
Acronym: Smart-screen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); Milpa Alta Municipalty (Unknown); Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government); Centro Interdisciplinario de Ciencias de la Salud, Mexico (Unknown); Educational Institutions of Milpa Alta (Unknown)
Responsible Party: Sponsor
Other Study IDs: SmartMexSurvey1
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Suicidal Ideation; Depression; Depressive Disorder; Anxiety; Alcohol Abuse; Drug Abuse
Keywords: Mass Screening; Health Surveys; Mental Health; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation; Depression; Depressive Disorder; Anxiety Disorders; Alcoholism; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Milpa Alta inhabitants: Population among 15 and 70 years old
  Interventions: Other: Self-administered evaluation questionnaire

INTERVENTIONS:
Other: Self-administered evaluation questionnaire — Smartphone app with MeMind questionnaires

SUMMARY:
The objective of this study is to make a suicide screening in the entire population of Milpa Alta (approximately 150,000 inhabitants), taking into account other outcomes such as depression, anxiety, alcohol and drugs. For this, an app for Smartphone (MeMind) or a web platform (www.MeMind.net) will be used in which the participants will take a self-administered questionnaire, composed of several psychometric instruments .

It is expected that 70% of the population between 15 and 70 years old can do so directly with their own Smartphone, although web access posts will be enabled in educational and municipal units to avoid discrimination based on age or access to technology.

Our main hypothesis argues that the early identification of people at risk in almost the entire community can be done with an App for Smartphone, serving to depict a map of mental health and related needs of the population, serving for the planning of healthcare services of the local environment, and ultimately for the best assistance of groups and individuals with greater needs through their identification and early reference to medical assistance.

ELIGIBILITY:
Inclusion Criteria:

1. Use a smartphone as personal or computer terminals enabled by the municipality of Milpa Alta or educational services.
2. Be able to understand the nature, purpose and methodology of the study.
3. Accept participation in the study and check the corresponding box in the app to verify that the informed consent has been expressly given.

Exclusion Criteria:

1. Subject deprived of liberty (by judicial or administrative decision)
2. Subject protected by law (guardianship or conservatorship)

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community composed of school population between 15 and 24 years of the educational institutions of Milpa Alta, and adult population of the municipality of Milpa Alta.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-01-23 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation | 1 Day
  Columbia-Suicide Severity Rating Scale (C-SSRS) is encompassed into MeMind for this purpose.
  In C-SSRS, four constructs are measured. The first is the severity of ideation, which is rated on a 5-point ordinal scale from 1="wish to be dead" to 5="suicidal intent with plan".
  The second is the intensity of ideation, which comprises 5 items, each rated on a 5-point ordinal scale: frequency, duration, controllability, deterrents, and reason for ideation.
  The third is the behavior, which is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
  And the fourth is the lethality, which assesses actual attempts; actual lethality is rated on a 6-point ordinal scale.
  Results are coded in the instrument itself with colored labels that indicates definitions of suicidal ideation and behavior, quantify both of them and gauge their severity.
  Definitions are available elsewhere (http://cssrs.columbia.edu).

SECONDARY OUTCOMES:
Depression | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to depression.
  PHQ-9 questionnaire is emcompassed into Memind for this purpose.
Anxiety | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to anxiety.
  GAD-7 (only screening questions) is emcompassed into Memind for this purpose.
Drug Utilization | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to anxiety.
  DAST (only questions 1,6,7) is emcompassed into Memind for this purpose.
Alcohol Drinking | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to alcohol abuse.
  Alcohol Use Disorders Identification Test (AUDIT-C)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcaldía Milpa Alta. Ciudad de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for researchers upon request
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Upon request to Enrique Baca Garcia (enrique.baca@uam.es)

REFERENCES:
- [Derived] Arenas-Castaneda PE, Aroca Bisquert F, Martinez-Nicolas I, Castillo Espindola LA, Barahona I, Maya-Hernandez C, Lavana Hernandez MM, Manrique Miron PC, Alvarado Barrera DG, Trevino Aguilar E, Barrios Nunez A, De Jesus Carlos G, Vildosola Garces A, Flores Mercado J, Barrigon ML, Artes A, de Leon S, Molina-Pizarro CA, Rosado Franco A, Perez-Rodriguez M, Courtet P, Martinez-Ales G, Baca-Garcia E. Universal mental health screening with a focus on suicidal behaviour using smartphones in a Mexican rural community: protocol for the SMART-SCREEN population-based survey. BMJ Open. 2020 Jul 19;10(7):e035041. doi: 10.1136/bmjopen-2019-035041. PMID 32690505
- See also: Related Info — http://www.MeMind.net